CLINICAL TRIAL: NCT07357662
Title: Evaluation of the Effects of Rehabilitative Exergame Exercises on Foot Muscle Activation, Balance, and Mobility in Older Adults Using Surface Electromyography and Postural Sway Measurements
Brief Title: Effects of Rehabilitative Exergame Training on Foot Muscle Activity, Balance, and Mobility in Older Adults
Acronym: EXG-FOOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Fatma Kübra ÇEKOK, Asst.prof, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tarsus U
Record Dates: First submitted 2026-01-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Aging; Foot Muscle Dysfunction; Sarcopenia; Age-Related Muscle Weakness
Keywords: older adults, physical activity, interactive computer games, biomarkers, electrophysiology, biomedical signal processing; Older adults; Biomedical signal processing; Physical activity
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame-based Balance and Foot Muscle Training (Experimental): Participants in the intervention group will undergo an 8-week supervised exercise program, consisting of 40-minute sessions performed two times per week. Each session will include a 5-minute warm-up, followed by the main exergame-based balance and foot muscle training, and a 5-minute cool-down period. The exercises will focus on improving postural control, foot muscle activation, balance, and mobility using rehabilitative exergame applications.
  Interventions: Other: Exergame-based Balance and Foot Muscle Training
- Functional balance training (Active Comparator): Participants in the control group will receive an 8-week supervised functional balance training program, consisting of 40-minute sessions performed two times per week. Each session will include a 5-minute warm-up, followed by 30 minutes of conventional functional balance exercises (such as static and dynamic standing balance, weight shifting, step training, and postural stabilization tasks), and a 5-minute cool-down period.
  Interventions: Other: Conventional Functional Balance Training

INTERVENTIONS:
Other: Exergame-based Balance and Foot Muscle Training — The interventions will carried out two days a week and 40 minutes, for eight weeks.
  Arms: Exergame-based Balance and Foot Muscle Training
Other: Conventional Functional Balance Training — he interventions will carried out two days a week and 40 minutes, for eight weeks.
  Arms: Functional balance training

SUMMARY:
This study is designed as a randomized controlled trial. A total of 40 healthy older adults residing in private and public nursing homes and rehabilitation centers in Mersin will be enrolled. Participants will be randomly assigned to either the intervention group (Group 1) or the control group (Group 2).

The intervention group will receive rehabilitative interactive game-based exercise training, while the control group will receive functional balance exercise training. Both groups will participate in exercise sessions three times per week, with each session lasting 40 minutes, over a period of 8 weeks.

Participants will undergo pre- and post-intervention assessments, including:

i) clinical tests and measurements for cognitive, functional, and balance evaluation; ii) surface electromyography (sEMG) measurements recorded during the Functional Reach Test (FRT); and iii) biomechanical measurements obtained via integrated inertial measurement unit (IMU) sensors (accelerometer and gyroscope) and the Becure game board.

Electrophysiological and biomechanical data will be analyzed using statistical comparisons, correlation analyses, and regression models. Variables derived from time, frequency, and time-frequency domain analyses will be examined to identify potential sEMG and biomechanical biomarkers.

DETAILED DESCRIPTION:
The increasing prevalence of sedentary lifestyles among older adults represents a major public health concern, as it accelerates age-related declines in physical mobility, muscle strength, postural control, and balance. These declines contribute to an increased risk of falls, highlighting the need for effective and innovative intervention strategies.

Rehabilitative interactive games (exergames) have emerged as a promising intervention by combining motor learning components, such as balance and functional mobility, with cognitive engagement. However, the effects of exergames on lower extremity functionality, balance performance, and their association with neuromuscular activity remain insufficiently understood.

This study adopts an innovative approach by employing surface electromyography (sEMG) to investigate electromyography-force relationships in trunk, leg, and foot muscles-an area that has received limited attention in the existing literature. While prior research has predominantly focused on traditional clinical assessments such as the Functional Reach Test (FRT) or ankle joint biomechanics, this study emphasizes the functional contribution of muscles involved in foot arch stabilization and toe control. This perspective aims to provide additional insight into the coordinated roles of foot, leg, and trunk musculature in balance and mobility.

The study will be conducted as a randomized controlled trial including 40 healthy older adults residing in nursing homes and rehabilitation centers in Mersin. Participants will be randomly allocated to either an intervention group receiving exergame-based exercise training or a control group receiving functional balance exercises. Both groups will complete 40-minute exercise sessions three times per week for a duration of eight weeks.

Pre- and post-intervention assessments will include:

i) clinical tests and measurements evaluating cognitive, functional, and balance performance; ii) surface EMG recordings obtained during the Functional Reach Test to assess muscle activity of the trunk, thigh, leg, and foot; and iii) biomechanical data collected using force plates and integrated IMU sensors (accelerometers and gyroscopes) synchronized with the surface EMG system.

Collected data will be analyzed across time, frequency, and time-frequency domains to examine relationships between electrophysiological and biomechanical variables. Statistical analyses will include comparative analyses, correlation analyses, and regression models to identify potential electrophysiological and biomechanical biomarkers associated with balance performance and exercise-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 to 80 years
* Having a minimum of 5 years of formal education
* Ability to walk independently for at least 10 meters, with or without a walking aid if necessary
* Having sufficient cognitive function for communication and participation, defined as a Mini-Mental State Examination (MMSE) score ≥26

Exclusion Criteria:

* Body mass index (BMI ≥30 kg/m²)
* Presence of central or peripheral nervous system disorders or use of medications that may affect balance
* History of vestibular pathology
* Lower extremity amputation, prior lower extremity surgery, or malignancy affecting the lower extremities
* Presence of moderate to severe congenital heart disease, coronary artery disease, or cerebrovascular disease
* Presence of visual, psychiatric, or cognitive impairments that could interfere with study participation or assessment procedures

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Standardized Mini-Mental State Examination (SMMSE). | Baseline (Pre-intervention assessment, Week 0)
  The Standardized Mini-Mental State Examination (SMMSE) is a widely used, brief cognitive screening tool adapted from the original Mini-Mental State Examination. It evaluates global cognitive function across several domains, including orientation, attention, immediate and delayed memory, language, and visuospatial abilities. The total score ranges from 0 to 30, with lower scores indicating greater cognitive impairment. The SMMSE is administered face-to-face and typically requires 5-10 minutes to complete. In this study, the SMMSE is used to screen cognitive eligibility and ensure participants have sufficient cognitive capacity to follow instructions and provide informed consent.
Surface EMG Frequency-Domain Parameters During Functional Reach Test | baseline and 8 weeks later
  Surface EMG Frequency-Domain Parameters During Functional Reach Test
  Description:
  Frequency-domain characteristics of the surface EMG signal will be analyzed during the Functional Reach Test to evaluate neuromuscular activation patterns. Parameters such as median frequency and mean frequency will be extracted to assess muscle activation characteristics.
  Unit of Measure:
  Hertz (Hz)
  Time Frame:
  Baseline (Week 0) and Post-intervention (Week 8)
Timed Up and Go Test (TUG) | Baseline (Week 0) and Post-intervention (8 Week )
  The Timed Up and Go (TUG) test is one of the most commonly used clinical tools for the assessment of balance and gait and is recommended by clinical practice guidelines for evaluating fall risk (Bohannon, 2006). This relatively simple assessment measures the time required for an individual to stand up from a chair, walk 3 meters, turn, return to the chair, and sit down, with the total duration recorded in seconds. A cut-off value of 14 seconds has been suggested to indicate increased fall risk.
  In the Cognitive Timed Up and Go test (TUG-cognitive), participants are additionally instructed to count backward by threes as quickly and safely as possible, starting from a randomly selected number between 20 and 100, while performing the motor task. A cognitive task duration of ≥15 seconds has been reported to predict backward falls with an accuracy of 87%.
Electrophysiological Measurements Using Surface EMG | Baseline (Week 0) and Post-intervention (Week 8)
  Surface EMG Muscle Activation During Functional Reach Test
  Description:
  Surface electromyography (sEMG) will be used to assess neuromuscular activation of trunk and lower extremity muscles during the Functional Reach Test. Muscle activation will be quantified using amplitude-based parameters derived from the sEMG signal, including root mean square (RMS) values.
  Unit of Measure:
  Microvolts (µV), RMS
  Time Frame:
  Baseline (Week 0) and Post-intervention (Week 8)
Center of Pressure (CoP) Displacement | Baseline (Week 0) and Post-intervention (Week 8)
  Center of pressure displacement will be measured using the Sensormedica platform to assess postural control. Anterior-posterior and medial-lateral CoP displacement will be analyzed during balance tasks.Unit of Measure:
  Millimeters (mm) or centimeters (cm)
Postural Sway Parameters | Baseline (Week 0) and Post-intervention (Week 8)
  Postural sway characteristics, including CoP path length and CoP velocity, will be assessed during static and dynamic balance tasks using the Sensormedica system.Unit of Measure:
  Centimeters (cm), centimeters per second (cm/s)
Lower Extremity Load Symmetry | Baseline (Week 0) and Post-intervention (Week 8)
  Load symmetry between the lower extremities will be evaluated during balance tasks using plantar pressure data obtained from the Sensormedica system.
  Unit of Measure:
  Percentage (%)

SECONDARY OUTCOMES:
Mini-Balance Evaluation Systems Test | Baseline (Week 0) and Post-intervention (Week 8)
  The Mini-Balance Evaluation Systems Test (Mini-BESTest) is a clinical assessment tool primarily focused on evaluating dynamic balance. It is widely used to assess balance impairment and fall risk. The scale consists of 14 task items, representing the four major balance control systems derived from the original BESTest: anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait stability.
  The test includes functional tasks such as standing, rising onto the toes, single-leg stance, forward, backward, and lateral reactive stepping responses, gait speed changes, head turns during walking, obstacle negotiation, and timed walking tasks performed on foam surfaces and inclined surfaces with eyes closed, as well as walking with changes in gait pattern. Higher scores indicate better dynamic balance performance.
Lower Extremity Muscle Strength (MicroFET 2 Handheld Dynamometer) | Baseline (Week 0) and Post-intervention (Week 8
  Lower extremity muscle strength in older adults will be assessed using the MicroFET 2 Handheld Dynamometer . Muscle strength is defined as the maximum voluntary isometric contraction (MVIC) achieved under standardized testing conditions. For each muscle group, participants will perform three maximal voluntary contractions. During each trial, force will be gradually increased over 2 seconds and then maintained at the maximal level for 3 seconds. The highest recorded value will be used for analysis.
  The following muscle groups will be tested:
  1. Knee extensor strength: Measured in the sitting position with the knee joint in extension.
  2. Knee flexor strength: Measured in the prone position with the knee joint in flexion.
  3. Ankle dorsiflexor strength: Measured in the sitting position with the ankle in dorsiflexion.
  4. Ankle plantar flexor strength: Measured in the sitting position with the ankle in plantar flexion.
Four Square Step Test (FSST) | Baseline (Week 0) and Post-intervention (Week 8)
  The test assesses dynamic balance. As a clinical assessment, it is reliable and valid in older adults, easy to administer and score, quick to perform, requires minimal space, and does not require specialized equipment. Owing to its evaluation of movement in four directions and the inclusion of low-height obstacles (2.5 cm), it is considered a unique assessment tool (Dite & Temple, 2002).

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma kübra çekok, Tarsus, Mersin, Turkey (Türkiye)